CLINICAL TRIAL: NCT03092492
Title: AMD Ryan Initiative Study
Brief Title: AMD Ryan Initiative Study (ARIS)
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170071; 17-EI-0071
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10-23

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Age-Related Macular Degeneration (AMD); Reticular Pseudodrusen; Natural History
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Participants with bilateral early AMD and medium drusen in both eyes
- Cohort 2A: Participants with at least one eye with RPD , with small or medium-sized drusen in either eye
- Cohort 2B: Participants with at least 1 eye with RPD, with large drusen in either eye
- Cohort 3: Healthy age-matched controls

SUMMARY:
Objective:

To learn more about AMD.

Eligibility:

People ages 55 and older with any of the following:

Early AMD

RPD

Healthy eyes

Design:

Participants will be screened with:

Eye exam: The pupil will be dilated with eye drops. Eye pressure and movements will be checked. Pictures will be taken of the inside of the eye.

Reading an eye chart.

Optical coherence tomography (OCT): The eyes are dilated. A machine measures the thickness of the retina.

Participants will have a first visit that includes:

Repeat of screening procedures

Medical history

Physical exam

Questions about vision and general health

Dark adapted fundus perimetry: Participants sit in the dark for 40 minutes. Then they sit at a machine that shines lights in the eyes.

Dark adaption testing: Participants sit in the dark for 45 minutes. The pupils are dilated. They push a button when they see light in a machine for up to 1 hour.

Participants will have annual visits for up to 5 years to repeat the tests in the first visit. Participant data may be shared for other research....

DETAILED DESCRIPTION:
Objective:

Late age-related macular degeneration (AMD) is the leading cause of blindness among elderly in the United States. At present, the current classification systems do not take into consideration advances in imaging technology, visual function biomarkers, as well as genotyping and phenotyping.

Clinical sites in the United States and around the world will conduct a longitudinal study that will bring together resources and commitment for the development of a classification scheme for AMD using imaging and visual function biomarkers, with the plan to correlate genetic information obtained in the future. These data could eventually help develop an understanding of the mechanisms involved in the development and progression of AMD. The project will recruit participants with early AMD or reticular pseudodrusen (RPD) and controls. All data and images from this longitudinal study will be available to researchers worldwide to help in the development of visual function biomarker identification and classification development. The initiative should provide an unparalleled state-of-the-art standardized phenotype and genotype including AMD status with information on imaging, visual function and biomarkers, with a particular focus to developing surrogate outcome variables for proof of principle phase 2 clinical trials.

Study Population:

This cohort study will recruit up to 500 total participants with early AMD or RPD, including age-matched controls.

Design:

This study is designed as a multi-center, international, prospective, observational cohort study of participants with early AMD or RPD. Study participants will undergo clinical assessments, multi-modal imaging and receive the standard of care as determined by the participant s ophthalmologist.

Outcome Measures:

Further research is necessary to characterize RPD and to understand the progression of AMD from early to late stage disease. The primary objectives of the longitudinal observational study are to enroll participants with early AMD (medium size drusen) to assess rate of change in drusen volume and progression rates to large drusen, and associate these morphologic changes with psychophysical changes, including visual acuity and dark adaptation. Separately, participants with RPD (verified by Reading Center review) will be enrolled and followed to better understand the natural history of RPD as well as to document structural and functional changes over time and associate them with the psychophysical changes listed above and changes in quality of life. In addition, control participants with no drusen or little drusen (normal aging changes) will be enrolled as comparison groups for the early AMD and reticular drusen groups. Data from this study will be analyzed to identify potential risk factors for disease progression and possible outcome variables for future studies. The collection of multi-model imaging at baseline and longitudinally will allow for an assessment of the disease classification and morphologic changes that might serve as biomarkers for disease progression for eyes with early AMD or RPD. Psychophysical testing will help assess functional changes and associations. Information will be disseminated to help the ophthalmic community better understand the natural course of early AMD and RPD.

To meet these objectives, the study will encourage up to approximately 20 sites participating in the AMD Ryan Initiative Study (ARIS) to recruit and characterize patients with early AMD or RPD for the longitudinal study.

The longitudinal phase of ARIS will collect information on consenting participants with early AMD or RPD seen at participating sites. Routine data collection will focus on the following:

* Enhancing the understanding of the natural history of early AMD and RPD
* Evaluating the functional characteristics of early AMD and RPD
* Compiling information on the potential ocular associations and natural progression of RPD
* Evaluating risk factors for disease progression in participants with early AMD and RPD
* Evaluating multi-model imaging to understand the mechanisms involved in the pathogenesis of early AMD and RPD
* Determining the 5-year progression rate to large drusen or late AMD in eyes with early AMD or RPD (in those participants who have NO large drusen at baseline)
* Determining the rate of change in drusen volume in eyes with early AMD and possibly the rate of change in the volume of sub-retinal deposits in eyes with RPD, stratified by the presence or absence of large drusen
* Compare the rates of progression in RPD in eyes with and without early or intermediate AMD
* Developing possible surrogate outcome variables associated with progression to late AMD or visual acuity loss including change in drusen volume
* Improving classification criteria for RPD

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in the longitudinal study, the potential participant must meet all of the following criteria.

* Men and women aged 55 and older;
* Clinical and Reading Center verification:

  * Cohort 1 - Early AMD, N=200 (Medium drusen >=63mu and <125mu) OU
  * Cohort 2 - RPD, N=200, (2A)At least one eye with RPD with no large drusen (>=125mu) in either eye; (2B)At least one eye with RPD with >=1 large drusen (>=125mu) in either eye (n=100)
  * Cohort 3 - Controls, N=100, No medium or large drusen, no peripheral drusen, no RPD or pigmentary changes OU
* Best Corrected Visual Acuity of 20/25 or better;
* Previous ocular surgeries allowed include cataract surgery more than three months prior to enrollment in ARIS and peripheral laser, cryotherapy for peripheral tears;
* Participant must be able to review and understand the informed consent form, agree to the contents and be able to sign the informed consent.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

* Any evidence of late AMD (i.e. CNV or GA) in either eye.
* Ocular disease other than AMD in either eye, in the Investigator's opinion, which may confound assessment of the retina including:

  * Amblyopia (in study eye only for Cohort 2)

    * Angioid streaks
    * Choroidal nevus within 2 DD of the center of the macula associated with depigmentation or overlying atypical drusen
    * Epiretinal membrane of significant size located in the macular area that potentially can cause vision loss
    * Myopic crescent of the optic disc the width of which is greater than or equal to 50% of the longest diameter of the disc, or pigmentary abnormalities in the posterior pole considered by the clinic ophthalmologist more likely to be due to myopia than to AMD
  * Central Serous Choroidopathy

    * Optic Atrophy
    * Diabetic retinopathy unless retinopathy is limited to fewer than 10 microaneurysms and/or small retinal hemorrhages
    * Macular hole or pseudohole
    * Pigmentary abnormalities considered by the Clinical Site ophthalmologist to be less typical of AMD than of some other condition, such as pattern dystrophy or chronic central serous retinopathy
  * Retinal vein occlusion, active uveitis, presumed ocular histoplasmosis syndrome, other sight-threatening retinopathies, and other retinal degenerations, significant explained or unexplained visual field loss, or any other type of retinopathy or retinal degeneration
* Previous retinal or other ocular surgical procedures, the effects of which may now or in the future complicate assessment of the progression of AMD in the Investigator s opinion;

  * These surgeries can be divided into those for 1) glaucoma: argon laser trabeculoplasty, trabeculectomy, and other penetrating glaucoma surgery involving valves, etc., 2) retinal diseases: laser photocoagulation (except to repair a peripheral retinal hole), cryosurgery (except any procedure to repair a peripheral retinal hole), intravitreal injections, vitrectomy 3) Refractive surgery:

Lasik, peripheral radial keratotomy (PRK), KAMRATM (corneal inlay for correction of presbyopia), 4) corneal diseases: lamellar keratoplasty, penetrating keratoplasty (PKP), Descement Membrane Endothelial Keratoplasty (DMEK), Descemet Stripping Endothelial Keratoplasty (DSEK), DSEK-A (DSEK-automated), Ultra-thin DESK, Deep Anterior lamellar Keratoplasty (DALK),

5) pterygium surgery that affects or threatens the visual axis, Others) radiation for ocular tumor, repair of corneal or sclera laceration.

* Retinal laser treatments and cryosurgery for retinal tears is not an exclusion.

  * Any other ocular condition requiring long-term therapy or surgery during the study or any other retinal pathology that in the Investigator s opinion will interfere with the interpretation of the macular AMD findings (e.g., CRVO);
  * Participants with confirmed glaucoma (visual field and/or disc/nerve fiber layer defects);
* Participants with a current IOP > 26, a history of the diagnosis of increased intraocular pressure, glaucoma, past or present use of medications to control intraocular pressure, or disc/nerve fiber layer defects suggestive of glaucoma can be eligible if the absence of a glaucomatous visual field defect can be documented by a normal Goldmann, Humphrey or Octopus perimetry test within six months prior to qualification.

  * Participant has photographically significant corneal or media opacities;
  * Participant has, in the opinion of the Investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments;
  * Participant is medically unable to comply with study procedures or follow-up visits.
  * Participation in research study involving treatment for AMD.

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at the NIH site will be recruited from the current patient population in our eye clinic as well as from new referrals from area clinics and practices.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Enroll participants with early AMD (medium size drusen) to assess rate of change in drusen volume and progression rates to large drusen, and associate these morphologic changes with psychophysical changes, including visual acuity and dark adapta... | 5 years
  The collection of multi-model imaging at baseline and longitudinally will allow for an assessment of the disease classification and morphologic changes that might serve as biomarkers for disease progression foreyes with early AMD or RPD. Psychophysical testing will help assess functional changes and associations.
Better understand the natural history of RPD as well as to document structural and functional changes over time and associate them with psychophysical changes and changes in quality of life. | 5 years
  The collection of multi-model imaging at baseline and longitudinally will allow for an assessment of the disease classification and morphologic changes that might serve as biomarkers for disease progression foreyes with early AMD or RPD. Psychophysical testing will help assess functional changes and associations.
Identify potential risk factors for disease progression and possible outcome variables for future studies | 5 years
  Data from this study will be analyzed to identify potential risk factors for disease progression and possible outcome variables for future studies. Information will be disseminated to help the ophthalmic community better understand the natural course of early AMD and RPD

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-EI-0071.html